CLINICAL TRIAL: NCT04939922
Title: China Headache and Vertigo Registry Study
Acronym: CHRS
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang University (Other); Tiantai People Hospital (Unknown); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); Huzhou Central Hospital (Other); The Affiliated Hospital of Hangzhou Normal University (Other); Xin Hua Hospital of Zhejiang Province (Other); The First People's Hospital of Huzhou (Other); Zhongshan Hospital Of Traditional Chinese Medicine (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Affiliated Wenling Hospital of Wenzhou Medical University (Other); Hangzhou Hospital of Traditional Chinese Medicine (Other); Jiaxing Hospital of T.C.M (Unknown); Shaoxing People's Hospital (Other); The First People Hospital of Hangzhou Lin An District (Unknown); The People's Hospital of Quzhou (Other); Affiliated Hospital of Jiaxing University (Other); First People's Hospital of Hangzhou (Other); SIR RUNRUN Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-0283
Record Dates: First submitted 2021-06-14; First posted 2021-06-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Headache Disorders, Primary; Headache Disorders, Secondary; Migraine; Tension-Type Headache; Cluster Headache; Vertigo, Constant; Vestibular Migraine; Fibromyalgia
Keywords: Migraine; Headache Disorders; Vertigo; Vestibular Migraine; Fibromyalgia
MeSH Terms: conditions — Headache Disorders, Primary; Headache Disorders, Secondary; Migraine Disorders; Tension-Type Headache; Cluster Headache; Vertigo; Fibromyalgia; Headache Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — Blood and urine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (5):
- Migraine: Patients with migraine (including vestibular migraine), including all types of migraine as defined by ICHD-3
- Other Primary Headache Disorders: Patients with other primary headache disorders (excluding migraine), including all types of other primary headache disorders (such as Tension-Type Headache, Cluster Headache) as defined by ICHD-3.
- Vertigo: Patients with other vertigo disorders (excluding vestibular migraine).
- Secondary Headache Disorders: Patients with secondary headache disorders as defined by ICHD-3.
- Normal control: Normal people do not have headache and vertigo.

SUMMARY:
In the Chinese Headache and Vertigo Registration Study, patients aged 4-99 years with headache (primary headache and secondary headache such as migraine and tension type headache), vertigo (vertigo diseases such as vestibular migraine) and chronic pain (fibromyalgia and other diseases) were collected. The biomarkers, imaging features, right-to-left shunt of the heart (lung), genetic characteristics, treatment, and outcome (in relation to other diseases) of headache-related diseases were studied, and long-term follow-up was planned.

DETAILED DESCRIPTION:
1. Research contents:

   In the Chinese Headache and Vertigo Registration Study, patients aged 4-99 years with headache (primary headache and secondary headache such as migraine and tension type headache), vertigo (vertigo diseases such as vestibular migraine) and chronic pain (fibromyalgia and other diseases) were collected. The biomarkers, imaging features, right-to-left shunt of the heart (lung), genetic characteristics, treatment, and outcome (in relation to other diseases) of headache-related diseases were studied, and long-term follow-up was planned.
2. Research target:

   We study biomarkers, imaging features, right-to-left shunt of heart (lung), genetic features, real-world treatment studies, and outcomes (in relation to other diseases) for headache and vertigo related diseases.
3. In order to ensure the quality of the trial, the sponsor and the researcher shall discuss and formulate the clinical research plan before the trial officially begins. GCP training was given to the relevant researchers who participated in the experiment. The research center must manage experimental drugs in accordance with (SOP), including receipt, storage, distribution and recycling. In accordance with the GCP guidelines, necessary steps should be taken during the design and implementation phase of the study to ensure that the data collected are accurate, consistent, complete and credible. All observed results and abnormal findings in clinical trials should be verified and recorded in time to ensure the reliability of the data. The instruments, equipment, reagents and standards used in various examination items in clinical trials should have strict quality standards and ensure that they work under normal conditions. The researcher inputs the information required by the program into the eCRF, and the inspector verifies whether the filling is complete and accurate, and instructs the staff of the research center to make necessary corrections and supplements. The drug regulatory department, the institutional review committee (IRB)

   / independent ethics committee (IEC), sponsor inspectors and / or inspectors may conduct systematic inspections of clinical trial-related activities and documents to evaluate whether trials are conducted in accordance with the requirements of the study program, SOP and relevant regulations (e.g. GCP, GMP), and whether trial data are recorded in a timely, true, accurate and complete manner. The inspection should be carried out by personnel who are not directly involved in the clinical trial. In order to meet the audit and / or inspection requirements of the regulator

   , the researcher / institution must agree to keep the relevant records, including the identification numbers of all subjects (sufficient information is linked to the records, such as eCRF and hospital records), all originally signed informed consent forms. All eCRF copies, safety report forms, original records, treatment details, related communication documents (such as letters, meeting minutes, phone reports). Researchers / institutions are required to keep records in accordance with relevant specifications.

   Relevant Chinese regulations and research institutions' requirements for the protection of subjects' personal information. Authorized representatives and regulatory agencies to examine (and copy if permitted by law) clinical records for quality review, inspection, and evaluation of safety, research progress and data validity. Raw data is all the information necessary to reconstruct and evaluate clinical research and is the original record of clinical findings, observations or other activities. Examples of these original documents and data records include, but are not limited to: hospital records, laboratory records, memos, subject diary cards, pharmacy dispensing records, audio recordings of consultation meetings, automated instrument records, verified as accurate and complete copies or transcripts, microfilm, photographic negatives, microfilms or disks, x-rays and stored in pharmacies participating in the study, documents and records of subjects in laboratories and medical technology departments.
4. Statistical analysis plan Differences between the two groups will be tested using the Mann-Whitney U test. P <0.05 indicates a significant difference. SPSS will be used. All statistical analyses will be based on the intent-to-treat principle using the full analysis set.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and participant privacy information (eg, Written Authorization for Use and Release of Health and Research Study Information) obtained from the participant prior to initiation of any study-specific procedures.
* Male or female participants ages 4 to 99 years.
* Headache patients meeting the diagnostic criteria for ICHD-3, including primary headaches such as migraine and tension tension-type headaches, secondary headaches.
* Patients who meet the headache diagnosis in the ICHD-3 appendix (including vestibular migraine).

Exclusion Criteria:

* Patients who were unable to complete scales such as headache diary.
* Patients denied or unable to be admitted for long-term follow-up.

Ages: 4 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Male or female participants ages 4 to 99 years
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-06-12 (Actual); Primary Completion 2050-12-12 (Estimated); Study Completion 2050-12-12 (Estimated)

PRIMARY OUTCOMES:
Days of Migraine | Medium term: within 6 months after initial diagnosis; long term: 30 years
  The number of days of migraine is the number of days in which migraine occurs or is likely to be migraine (according to IHS ICHD-3 diagnostic criteria).
  A migraine day is a day when a headache lasts for more than 30 minutes, does not take painkillers, and meets the ICHD-3 migraine or most likely migraine criteria. Migraine day can also be defined as a headache day that is effective for the acute treatment of specific migraine drugs (triptan, ditan, gepant, ergotamine, etc.).
Moderate / Severe Headache Days | Medium term: within 6 months after initial diagnosis; long term: 30 years
  Moderate / severe headache days are defined as a day in which moderate or severe pain persists for at least 4 hours, or headache lasts for one day after successful medication for acute headache. These definitions allow the use of relatively simple headache diaries. Subjects were required to indicate whether headache was present (yes / no), peak (mild / moderate / severe) severity and duration (< 4h or 4h), type of acute drug intake (triptan ergot / other), and response to treatment should also be recorded.
Vertigo attack | Medium term: within 6 months after initial diagnosis; long term: 30 years
  Vertigo is a sensation of feeling off balance. Vertigo attack is defined as any vertigo or dizziness attacks, such as the condition where person has the sensation of moving or of surrounding objects moving when they are not. Some questionnaires, such as the dizziness handicap inventory (DHI) and Vertigo Symptom Scale (VSS) are used to assess the severity of vertigo. The differential diagnosis of vertigo or dizziness can be narrowed with easy-to-perform physical examination tests, including evaluation for nystagmus, the Dix Hallpike maneuver, and orthostatic blood pressure testing.

SECONDARY OUTCOMES:
Migraine Attack | Medium term: within 6 months after initial diagnosis; long term: 30 years
  Migraine attack is defined as any consistent migraine attacks or the use of specific migraine drugs. If a migraine attack is interrupted by sleep, or temporarily relieved, and then relapses within 48 hours, it is considered an attack. In addition, migraine attacks that were successfully treated with drugs but relapsed within 48 hours and lasted for more than 48 hours were counted as one attack.
The Response Rate of at Least 50%, 75% and 100% Reduction in the Number of Days of Migraine Attacks | Medium term: within 6 months after initial diagnosis; long term: 30 years
  The response rate is calculated as the percentage reduction in the frequency of migraine attacks (or days of migraine, or days of moderate or severe headache) compared with the baseline during each treatment period. The response rate is traditionally defined as a reduction of at least 50% from the baseline, but other percentage reductions (for example: 30%, 75%, 100%) may be used.
Headache Intensity | Medium term: within 6 months after initial diagnosis; long term: 30 years
  Four-point rating scale was used to evaluate the headache intensity of each migraine day--painless, mild, moderate, or severe. Migraine intensity is not recommended as the main outcome measure alone, but it is important to record the decrease in migraine intensity as an indicator of disability reduction.
  Depending on the design of the trial, subjects should be asked to record the intensity of each migraine. In addition, the 11 point visual rating scale (VAS) can be used instead or in combination with the 4-level classification rating scale. The use of VAS in clinical trials may increase the likelihood of showing differences in severity.
Cumulative Hours of Moderate / Severe Pain | Medium term: within 6 months after initial diagnosis; long term: 30 years
  The cumulative number of hours of moderate / severe pain calculated by electronic headache diaries. If an attack occurs before going to bed and when you wake up, the amount of sleep also counts as the number of headache hours.
Days Without Symptoms | Medium term: within 6 months after initial diagnosis; long term: 30 years
  Defined as the number of days without aura, prodromal symptoms, headaches, pain and subsequent symptoms. It needs to be determined by headache diary.
Days Without Headache | Medium term: within 6 months after initial diagnosis; long term: 30 years
  The number of days without headache also includes the number of days without related symptoms directly caused by migraine (including physical function, cognitive or emotional disorders).
Peak Headache Pain Intensity | Medium term: within 6 months after initial diagnosis; long term: 30 years
  Subjects should record the maximum intensity of daily headaches and any medication used. An 11-point digital rating scale can be used instead of or in conjunction with a 4-level classified rating scale.
Acute Medication Use Day | Medium term: within 6 months after initial diagnosis; long term: 30 years
  An acute medication use day is defined as any day on which a participant reports, per eDiary, the intake of allowed medication(s) to treat an acute migraine. The allowed medications include the following categories of drugs: triptans, ergots, opioids, analgesics (including acetaminophen), NSAIDs (including aspirin), and antiemetics.
Activity Impairment in Migraine - Diary (AIM-D) | Medium term: within 6 months after initial diagnosis; long term: 30 years
  The AIM-D is a 9-item PRO measure that assesses the impact of migraine on the performance of daily activities and physical impairment. Participants are asked to rate the level of difficulty experienced in the past 24 hours with performance of daily activities (ie, difficulty with household chores, errands, leisure activities at home, leisure or social activities outside the home, strenuous physical activities) and physical impairment (ie, difficulty walking, moving body, bending forward, moving head) using a 6-point rating scale
Patient Difficulty in Concentrating, Difficulty in Thinking Clearly, Activity Level, and Activity Limitation | Medium term: within 6 months after initial diagnosis; long term: 30 years
  Four items based on a 24-hour recall will be administered daily using Headache and Non-Headache versions as additional health outcome measures and for evaluation of the AIM-D.
  The first item will be used to assess difficulty in concentrating with 6 responses ranging from "Not difficult at all" to "Extremely difficult" and an option of "I could not do it at all." The second item will be used to assess difficulty in thinking clearly with 6 responses ranging from "Not difficult at all" to "Extremely difficult" and an option of "I could not do it at all." The third item will be used to assess activity level within the past 24 hours with a 5-level response ranging from "No activity - Spent all day lying down" to "Exercised - Brisk walk, running, jogging, biking or other activity for 30 or more minutes." The fourth item will be used to evaluate activity limitation with a 5-level response ranging from "Not at all limited - I could do everything" to "Extremely limited."
Headache Impact Test (HIT-6) | Medium term: within 6 months after initial diagnosis; long term: 30 years
  The HIT-6 is a 6-question assessment used to measure the impact headaches have on a participant's ability to function on the job, at school, at home, and in social situations. It assesses the effect that headaches have on normal daily life and the participant's ability to function.
  Responses are based on frequency using a 5-point scale ranging from "never" to "always." The HIT-6 total score, which ranges from 36 to 78, is the sum of the responses - each of which is assigned a score ranging from 6 points (never) to 13 points (always).
Migraine Disability Assessment (MIDAS) | Medium term: within 6 months after initial diagnosis; long term: 30 years
  The MIDAS is a 7-item questionnaire designed to quantify headache-related disability over a 3- month period. The MIDAS score is the sum of missed work or school days, days at work or school plus days of household work where productivity was reduced by half or more, missed household work days, and missed non-work activity days due to headaches in the last 3 months.
Patient Global Impression of Change (PGIC) | Medium term: within 6 months after initial diagnosis; long term: 30 years
  The PGIC is a single item questionnaire used to measure the participant's impression of overall change in migraine since the first dose of study medication. The measure uses a 7-point rating scale with responses ranging from "very much better" to "very much worse."
Work Productivity and Activity Impairment Questionnaire Migraine V2.0 (WPAI:MIGRAINE) | Medium term: within 6 months after initial diagnosis; long term: 30 years
  The WPAI:MIGRAINE will be used to assess work productivity specific to migraine. The measure uses a 1-week recall and contains 6 questions related to work productivity. The WPAI measures both presenteeism and absenteeism. The measure yields four scores expressed as impairment percentages ranging from 0 to 100%: Percent work time missed, percent impairment while working, percent overall work impairment, and percent activity impairment due to migraine.
European Quality of Life - 5 Dimensional (EQ-5D-5L) | Medium term: within 6 months after initial diagnosis; long term: 30 years
  EQ-5D-5L is a generic instrument for use as a measure of health status. The EQ-5D-5L consists of 2 components - the EQ-5D descriptive system and the EQ VAS. The descriptive system comprises of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). The respondent is asked to indicate his/her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions.
  The scoring range of the EQ-5D descriptive system is typically from 0 (dead) to 1 (full health).
  The EQ VAS records the respondent's self-rated health on a vertical, VAS where the endpoints are labelled "Best imaginable health state" and "Worst imaginable health state." The scoring range of the EQ VAS is from 0 (worst imaginable health) to 100 (best imaginable health).
Patient Global Impression - Severity (PGI-S) | Medium term: within 6 months after initial diagnosis; long term: 30 years
  The PGI-S is a single item questionnaire used to measure the participant's impression of severity in relation to migraine symptoms overall at the time of administration of the measure. The measure uses a 5-point rating scale with responses ranging from "none" to "very severe."
Migraine Specific Quality of Life Questionnaire, Version 2.1 (MSQ v2.1) | Medium term: within 6 months after initial diagnosis; long term: 30 years
  The MSQ v2.1 is a 14-item questionnaire designed to measure health-related quality-of-life impairments attributed to migraine in the past 4 weeks. It is divided into 3 domains: Role Function Restrictive assesses how migraines limit one's daily social and work-related activities; Role Function Preventive assesses how migraines prevent these activities; and the Emotional Function domain assesses the emotions associated with migraines. Participants respond to items using a 6-point scale ranging from "none of the time" to "all of the time." Raw dimension scores are computed as a sum of item responses and rescaled to a 0 to 100 scale, where higher scores indicate better quality of life.
Patient-Reported Outcomes Measurement Information System Pain Interference - Short Form 6a (PROMIS-PI) | Medium term: within 6 months after initial diagnosis; long term: 30 years
  The PROMIS-PI measures self-reported interference of pain on relevant aspects of daily life (ie, social, cognitive, emotional, physical, recreational) over the past 7 days. A 5-level response scale for all six items ranges from "Not at all" to "Very much." Scores range from 6 to 30, with higher scores indicating greater pain interference.
Columbia-Suicide Severity Rating Scale | Medium term: within 6 months after initial diagnosis; long term: 30 years
  Suicidal ideation should be monitored in trials of central action drugs, higher scores mean a worse outcome.
  Many migraine clinical trials used the Columbia suicide severity scale (C SSRS).The C-SSRS consists of a maximum of 20 items. C-SSRS will be administered in study subjects at each study visit to assess possible suicidal ideation and behavior. Reports of suicidal ideation with intent to act (endorse item 4 or 5) and reports of actual, aborted, or interrupted suicide attempts or a behavior preparatory for making an attempt indicate subjects at high risk for suicide.
Generalized Anxiety Disorder (GAD-7) | Medium term: within 6 months after initial diagnosis; long term: 30 years
  GAD-7 is a proven, self-administered and concise tool for screening and diagnosing mental health disorders, which has been tested in the field in office practice. The screening scale is easy to use and can be completed in a short time, which improves the recognition rate of anxiety disorders and facilitates diagnosis and treatment. The main statistical index of this scale is the total score, that is, the sum of item scores. The total score range of GAD-7 is 0: 21 and that of GAD-2 is 0: 6. The score of GAD-7 can be used to evaluate the severity of anxiety symptoms: 0: 4: no clinical significance: anxiety: 5: 9: mild; 10: 14: moderate; > 15: severe. When used as an assistant diagnosis of anxiety symptoms, the cut-off value of GAD-7 is greater than or equal to 10.
Functional Impairment Scale (FIS) | Medium term: within 6 months after initial diagnosis; long term: 30 years
  Functional impairment scale (FIS) is a 4-point scale to evaluate the functional status and injury intensity in daily activities. It can be used in conjunction with the four-point pain intensity scale, usually done daily and summarized within four weeks.
Migraine Physiological Function Influence Diary (MPFID) | Medium term: within 6 months after initial diagnosis; long term: 30 years
  Migraine physiological function influence diary (MPFID) assessed the effect of migraine time during and between attacks on daily behavior and work.
Biomarkers of primary headache and vertigo | Medium term: within 6 months after initial diagnosis; long term: 30 years
  Blood samples will be collected from all participants who consent to participate in the substudy, for the purposes for future biomedical research, such as biomarkers of primary headache, such as inflammatory cytokines, neuropeptides and proteins.
Safety Measures, Adverse Events and Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Medium term: within 6 months after initial diagnosis; long term: 30 years
  Subjective AEs will be collected from the time of consent through the last visit. For all AEs, the investigator must provide an assessment of the severity, causal relationship to the investigational product, start and stop date, and seriousness of the event (eg, SAE), document all actions taken with regard to the investigational product, and detail any other treatment measures taken for the AE. For events noted as SAEs, Allergan must be notified immediately to meet their reporting obligations to appropriate regulatory authorities. Number of participants with treatment-related adverse events are assessed by CTCAE v4.0
Physical Examination | Medium term: within 6 months after initial diagnosis; long term: 30 years
  A complete physical examination (PE) per standard of care (including neurological exam) will be performed on all subjects. Any clinically significant anomalies noted during the initial screening phase are to be detailed in the Medical History CRF. Investigators are to check for any findings that would constitute study exclusion.
Medical and Medication History | Medium term: within 6 months after initial diagnosis; long term: 30 years
  A review of medical and medication history will be performed at initial screening to confirm subject eligibility. Targeted medical history is to be recorded in the Neurologic Medical History CRF and Cardiovascular Medical History CRF, and other medical history is to be recorded in the General Medical History CRF. Source notes for subjects referred to the research site must include all of the above information.
Physical Measurements | Medium term: within 6 months after initial diagnosis; long term: 30 years
  The following measurements are to be performed: height (initial screening only) and weight. Height and weight are to be measured without shoes. Body Mass Index (BMI) should be calculated using the following formula: BMI (kg/m2
  * = weight (kg)/[height (cm)/100]2
  All measurements are to be recorded on the Physical Measurements CRF.
Genetic analysis of familial headache and vertigo | Medium term: within 6 months after initial diagnosis; long term: 30 years
  Blood samples will be collected from all participants who consent to participate in the substudy, for the purposes for genetic analysis of familial headache and vertigo.disease.

CONTACTS AND LOCATIONS:
Overall Officials: Kaiming Liu, Doctor, Principal Investigator — headache specialist clinic of the Second Affiliated Hospital of Zhejiang Medical University
Locations (1):
- Kaiming Liu, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zou X, He J, Zhou M, Zhao F, Tian X, Xu X, Hong W, Wang F, Chen J, Qin C, Xia J, Xie Y, Xiao Y, Liu K, Guo L. Photophobia and Visual Triggers in Vestibular Migraine. Neurol Ther. 2024 Aug;13(4):1191-1201. doi: 10.1007/s40120-024-00631-8. Epub 2024 May 31. PMID 38819614
- [Derived] Xu X, Zhou M, Wu X, Zhao F, Luo X, Li K, Zeng Q, He J, Cheng H, Guan X, Huang P, Zhang M, Liu K. Increased iron deposition in nucleus accumbens associated with disease progression and chronicity in migraine. BMC Med. 2023 Apr 7;21(1):136. doi: 10.1186/s12916-023-02855-1. PMID 37024948
- [Derived] Liu K, Tian X, Hong W, Xiao Y, Chen J, Jin H, Wang F, Xu X, Zang T, Zhang L, Pan M, Zou X. Positive Relationship Between Paroxysmal Vertigo and Right-to-Left Shunt: A Large Observational Study. Front Neurol. 2022 Jun 3;13:927853. doi: 10.3389/fneur.2022.927853. eCollection 2022. PMID 35720061